CLINICAL TRIAL: NCT00019474
Title: Phase II Trial of 2-Fluorouracil Recombinant Alpha-2a-Interferon and Intravenous Hydroxyurea With Filgrastim in Patients With Refractory GI Malignancies Grant Application Title: Parenteral Hydroxyurea: A Modulator in Pancreatic Cancer
Brief Title: Combination Chemotherapy Plus Interferon Alfa Followed by Filgrastim in Treating Patients With Gastrointestinal Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066253; P30CA013330 (NIH); AECM-9707254; MMC-9007262-PHII; MMC-FDR001009-PHII
Record Dates: First submitted 2001-07-11; First posted 2004-04-13 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Extrahepatic Bile Duct Cancer; Gastric Cancer; Gastrointestinal Carcinoid Tumor; Liver Cancer; Pancreatic Cancer; Small Intestine Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; regional gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; small intestine adenocarcinoma; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; adult primary hepatocellular carcinoma; stage IV pancreatic cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Stomach Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Carcinoma, Hepatocellular | interventions — Filgrastim; Interferon-alpha; Fluorouracil; Hydroxyurea

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: fluorouracil
Drug: hydroxyurea

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person recover from the side effects of chemotherapy. Combining chemotherapy with interferon alfa may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy and interferon alfa followed by filgrastim in treating patients who have gastrointestinal tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rates in patients with unresectable locally advanced or advanced gastrointestinal malignancy treated with intravenous hydroxyurea, fluorouracil, interferon alfa, and filgrastim (G-CSF). II. Determine the toxic effects of this regimen in these patients. III. Determine the reversal of toxic effects of this regimen in these patients.

OUTLINE: Patients are stratified according to site of primary disease (hepatobiliary vs gastric vs pancreatic). Patients receive fluorouracil IV over 48 hours and hydroxyurea IV over 48 hours on days 1, 8, 22, and 29. Patients also receive interferon alfa subcutaneously (SC) on days 1, 3, and 5 and filgrastim (G-CSF) SC on days 3-6 of weeks 1, 2, 4, and 5. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 31-60 patients (18-33 with hepatobiliary or gastric cancer and 13-27 with pancreatic cancer) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed pancreatic, gastric, biliary system, or hepatocellular carcinoma beyond the scope of surgical resection Gastrointestinal tract carcinoid tumor or carcinoma of the small bowel allowed Bidimensionally measurable disease Ineligible for ECOG 6296 (gastric cancer) No brain metastases, unless completely resected and CT scan of the brain is normal

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 3 times normal SGOT less than 3 times normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease No chronic or uncontrolled angina No significant coronary artery disease (even if asymptomatic) on cardiac catheterization or thallium stress test, in patients with a history of atherosclerotic heart disease No congestive heart failure No arrhythmia Pulmonary: No chronic obstructive pulmonary disease No chronic pulmonary disease, including asthma, chronic bronchitis, emphysema, sarcoid, or bronchiectasis Neurologic: No cerebellar disease No seizure disorder Other: HIV negative No active or serious underlying infection No AIDS No psychiatric illness No organic mental syndrome No major psychoaffective disorder No poorly controlled diabetes mellitus No serious underlying illness that would preclude study No recent history of alcohol or drug abuse Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No prior systemic chemotherapy for advanced disease Prior fluorouracil or gemcitabine as radiosensitizer allowed No other prior chemotherapy Endocrine therapy: No concurrent systemic steroids No concurrent hormonal therapy (excluding birth control pills) No concurrent steroids as antiemetics or for chronic treatment Radiotherapy: At least 1 month since prior radiotherapy Surgery: See Disease Characteristics Recovered from prior surgery Other: At least 1 week since prior beta blockers No concurrent chronic treatment with aspirin, non-steroidal anti-inflammatory drugs, antihistamines, antianginal medication, extraordinary antihypertensive regimens, or antiarrhythmics (except cardiac glycosides)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1998-03; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wadler, MD, Study Chair — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Comprehensive Cancer Center, The Bronx, New York, United States